CLINICAL TRIAL: NCT06350279
Title: A Single and Multiple Ascending Dose Study to Assess the Safety,Tolerability, PK, PD, and Food Effect of HSK39297 in Healthy Subjects
Brief Title: A Phase I Study to Assess the Safety,Tolerability, PK, PD, and Food Effect of HSK39297 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HSK39297-101
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: HSK39297; healthy subjects; Phase I

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HSK39297 (Experimental): Single or multiple oral doses of HSK39297
  Interventions: Drug: HSK39297
- Placebo (Experimental): Placebo
  Interventions: Drug: HSK39297

INTERVENTIONS:
Drug: HSK39297 — 50-600mg

SUMMARY:
This is a Phase I, randomized, subject-blinded, placebo controlled study to assess the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD),and food effect (FE) of HSK39297 following (1) a single ascending dose (part 1), (2) 10 days of multiple ascending dose (part 2), and (3) a single dose two-period crossover FE cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form, understand the trialprocedures, and be willing to comply with all trial procedures andrestrictions;
2. 18 years to 45 years (inclusive), male and female;
3. Male subjects weight ≥50 kg and female subjects weight ≥45 kg. Bodymass index (BMI) : 18-26 kg/m2 (inclusive) ;
4. Subjects are willing to voluntarily use effectivecontraceptives from screening to at least 3 months after the last dose administration.

Exclusion Criteria:

1. Have a history of severe and uncontrolled diseases, such ascardiovascular, respiratory, liver, gastrointestinal, endocrine,hematologic, mental/nervous systems diseases within 3 months prior to screening;
2. Have an infection that requires systematic treatment with antibiotics, antifungal, antiparasitic or antiviral drugs;
3. Have a clear history of capsular bacteria infection within 6 months before screening, inncluding but not limited to Neisseria meningitidis, Streptococcus pneumoniae, Haemophilus influenzae B, etc.;
4. Have a history of TB infection or are currently infected with TB;
5. Have a history of any malignant tumors;
6. The abnormalities were clinically significant during the screening period, such as physical examination, vital signs, blood biochemistry, blood routine, coagulation, urine routine, blood pregnancy test, infectious diseases and X-ray;
7. Subjects whose results of routine 12-lead electrocardiograms were inconsistent with normal heart conduction and function;
8. Previous or current gastrointestinal, liver, kidney, or other disease known to interfere with drug absorption, distribution, metabolism, or excretion;
9. Smoking more than 5 cigarettes per day within 3 months prior toscreening or smoking during the study;
10. Average alcohol intake is more than 14 unit per week (1unit=10g alcohol , 1 unit=285 mL 4.9% alcohol beer, or 30 mL 40% alcohol spirit, or 100mL 12% alcohol wine) within the 3 months prior to screening;
11. Have a history of drug abuse prior to screening, or positive urine drug screen at screening;
12. Have a history of high consumption of grapefruit juice, methylxanthinerich food or beverage (such as coffee, tea, cola, chocolate, energydrinks) ,consumption of grapefruit juice, methylxanthine-rich food within 48 hours before the administration;
13. Blood donation (or blood loss) ≥400 mL, or receiving blood products to improve anemia within 3 months prior to the screening;
14. Subjects who have a allergic to any component of HSK30297 or allergic history to opiates;
15. Any drug that inhibits or induces drug metabolism enzymes or P-gp inhibitor have been administered within 28 days prior to initial administration of the investigational drug;
16. Subjects who use any live vaccine within 30 days prior to screening;
17. Have participated in any clinical investigator within 3 months prior to screening;
18. A pregnant/lactating woman, or has a positive pregnancy test at screening or during the trial;
19. Not suitable for this study as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) . | 9 days after single dose and 16 days after the first dose of multiple doses
  To assess the safety and tolerability of single or multiple oral dose of HSK39297 in healthy adult volunteers

SECONDARY OUTCOMES:
AUC | Pre-dose to 168 hours post-dose
  Area under the plasma concentration versus time curve (AUC) on Day 1 and D10
Cmax | Pre-dose to 168 hours post-dose
  The maximun plasma concentration of HSK39297
Tmax | Pre-dose to 168 hours post-dose
  Time of maximum concentration of HSK39297
t1/2 | Pre-dose to 168 hours post-dose
  half-life
AP change | Pre-dose to 168 hours post-dose
  change from baselin of the alternative pathway activity
Bb | Pre-dose to 168 hours post-dose
  change from baselin of the concentration of Bb

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No